CLINICAL TRIAL: NCT00873873
Title: Progression of Airway Obstruction in Childhood Asthma
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 645; R21HL087811-01 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: Asthma Progression; Airway Wall Thickness; Corticosteroid Resistance; Biomarkers; Pulmonary Physiology
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Induced sputum, urine, blood, and exhaled breath condensates
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Persistent obstruction: (pattern of asthma progression)
- Late obstruction: (pattern of asthma progression)
- Late normal: (pattern of asthma progression)
- Persistent normal: (pattern of asthma progression)

SUMMARY:
Distinct patterns of loss in pulmonary function were identified in children with mild to moderate asthma participating in a 10-year observation period during the NHLBI Childhood Asthma Management Program. This loss in pulmonary function is likely related to ongoing inflammation unresponsive to current therapy. This study will measure indicators of airway inflammation which are associated with structural and physiologic changes in the lung and provide insight into mechanisms of asthma progression in adolescence and early adulthood.

DETAILED DESCRIPTION:
The Childhood Asthma Management Program Continuation Study/Phase 2 is a 3.25 year observational follow-up study of the children enrolled in the Childhood Asthma Management Program (CAMP) randomized trial. CAMPCS/2 is a multicenter National Heart, Lung and Blood Institute program. The objective of the CAMPCS/2 is to determine the consequences of childhood asthma and its treatment on asthma outcomes in young adulthood. This separate ancillary study will extend the core CAMP/CAMPCS work by focusing on progression of airway obstruction in childhood asthma to evaluate mechanisms of progression and describe the differences in the four separate patterns in airway obstruction that have evolved over time. The four patterns of airway obstruction which have been identified are as follows: (1) abnormal obstruction present in early childhood which remained abnormal (Low/Low group) and (2) initially normal ratios, which worsened into the abnormal range over time (Normal/Low group). These patterns with unfavorable outcomes can be compared to two other patterns with favorable outcomes: (3) initially abnormal ratios improving with time (Low/Normal group) and (4) normal ratios throughout follow-up (Normal/Normal group).

Based on these four patterns, three specific hypotheses related to immunology, structure, and physiology are identified:

1. Among school-aged children with mild to moderate asthma, those children with increased airflow limitation (i.e. low FEV1/FVC) at the end of CAMPCS (Normal/Low and Low/Low groups) have elevated markers of inflammation related to proteolysis (i.e. neutrophil elastase, matrix metalloproteinase-9 (MMP9), and tissue inhibitor of metalloproteinase-1 (TIMP1) and neutrophils in sputum).
2. Subjects who show a pattern of early progression and failure to resolve (Low/Low group) have clinical evidence of steroid insensitivity compared to those with slow progression (Normal/Low group). They also have in vitro evidence of steroid resistance compared to the Normal/Low or Normal/Normal groups. This pattern of obstruction may be due to irreversible changes consistent with airway remodeling and inflammation that are relatively refractory to steroid therapy.
3. Children with ongoing airflow limitation (Normal/Low and Low/Low groups) have more prominent structural changes related to increased air trapping and airway thickening compared to those with normal FEV1/FVC at the end of CAMPCS (Low/Normal and Normal/Normal groups).

Each participant will be studied at varying times over the 2-year study period. Researchers will complete a collection of sputum, blood, urine, and exhaled breath condensate samples; exhaled nitric oxide; and spirometry from CAMPCS/3 participants, representing each of the four phenotypes (n = 20 for a total of 80).

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in the CAMPCS/3 study; individuals enrolled in this study will represent four different patterns of asthma progression, as defined by forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) levels

Exclusion Criteria:

* Unwilling to comply with study procedures
* Physical state does not allow the study procedures to be performed (e.g., low pulmonary function for induced sputum, pregnancy for computerized tomography [CT] scan)

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants enrolled in CAMPCS/3 from various CAMP sites will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J. Szefler, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Childhood Asthma Management Program Research Group; Szefler S, Weiss S, Tonascia J, Adkinson NF, Bender B, Cherniack R, Donithan M, Kelly HW, Reisman J, Shapiro GG, Sternberg AL, Strunk R, Taggart V, Van Natta M, Wise R, Wu M, Zeiger R. Long-term effects of budesonide or nedocromil in children with asthma. N Engl J Med. 2000 Oct 12;343(15):1054-63. doi: 10.1056/NEJM200010123431501. PMID 11027739
- [Background] Covar RA, Spahn JD, Murphy JR, Szefler SJ; Childhood Asthma Management Program Research Group. Progression of asthma measured by lung function in the childhood asthma management program. Am J Respir Crit Care Med. 2004 Aug 1;170(3):234-41. doi: 10.1164/rccm.200308-1174OC. Epub 2004 Mar 17. PMID 15028558
- [Background] Strunk RC, Weiss ST, Yates KP, Tonascia J, Zeiger RS, Szefler SJ; CAMP Research Group. Mild to moderate asthma affects lung growth in children and adolescents. J Allergy Clin Immunol. 2006 Nov;118(5):1040-7. doi: 10.1016/j.jaci.2006.07.053. PMID 17088127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The NHLBI Childhood Asthma Management Program (CAMP) and CAMP Continuation Studies afforded a unique opportunity to investigate four newly described, distinct patterns of airway obstruction associated with childhood asthma, including two that have been associated with significant and potentially irreversible loss in pulmonary function.
Pre-assignment Details: Analysis of serial pulmonary function measures in participants in CAMP and CAMPCS over time showed 4 patterns of airway obstruction developing during childhood and adolescence based on measurements of pre-bronchodilator FEV1/FVC at the time of enrollment in CAMP and again at the end of the observational phase.
Groups:
- Persistent Obstruction: This group represents those that have persistent obstruction from baseline at entry into the NHLBI CAMP study until end of the CAMP Continuation study, 9 years later.
- Late Obstruction in Pulmonary Physiology: This group represents those that had normal pulmonary function from baseline at entry into the NHLBI CAMP study and then has evidence of obstruction, as defined by FEV1/FVC criteria, at end of the CAMP Continuation study, 9 years later.
- Late Normal in Pulmonary Physiology: This group represents those that has evidence of obstruction, as defined by FEV1/FVC criteria, from baseline at entry into the NHLBI CAMP study and then has normal pulmonary function at end of the CAMP.
- Persistent Normal in Pulmonary Physiology: This groups has normal pulmonary function at the time of entry into the CAMP study and normal pulmonary function 9 years later.
Period: Overall Study
Arm/Group | Persistent Obstruction | Late Obstruction in Pulmonary Physiology | Late Normal in Pulmonary Physiology | Persistent Normal in Pulmonary Physiology
Started | 20 | 8 | 9 | 18
Completed | 20 | 8 | 9 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Persistent Obstruction | Late Obstruction in Pulmonary Physiology | Late Normal in Pulmonary Physiology | Persistent Normal in Pulmonary Physiology | Total
Number analyzed (Participants) | 20 | 8 | 9 | 18 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 1 | 3 | 9
  Between 18 and 65 years | 17 | 6 | 8 | 15 | 46
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (2.1) | 18.9 (2.0) | 20.8 (2.4) | 19.9 (2.0) | 20.0 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 6 | 11 | 27
  Male | 12 | 6 | 3 | 7 | 28
Region of Enrollment [Number; unit: participants]
  United States | 20 | 8 | 9 | 18 | 55

OUTCOME MEASURES:

1. Primary Outcome: Airway Wall Thickness
Description: Segmental average airway wall thickness
Time Frame: Measured at Year 2
Population: There were 43 participants with Chest CT data; 1 was excluded from the analysis due to incidental finding of an anatomical congenital anomaly.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Late Obstruction: This group represents those that had normal pulmonary function from baseline at entry into the NHLBI CAMP study and then has evidence of obstruction, as defined by FEV1/FVC criteria, at end of the CAMP Continuation study, 9 years later.
- Late Normal: This group represents those that has evidence of obstruction, as defined by FEV1/FVC criteria, from baseline at entry into the NHLBI CAMP study and then has normal pulmonary function at end of the CAMP.
- Persistent Normal: This groups has normal pulmonary function at the time of entry into the CAMP study and normal pulmonary function 9 years later.
Arm/Group | Persistent Obstruction | Late Obstruction | Late Normal | Persistent Normal
Number analyzed (Participants) | 15 | 7 | 8 | 12
mm | 1.5 (0.2) | 1.5 (0.2) | 1.4 (0.1) | 1.6 (0.3)
Statistical Analysis 1: Comparison: Persistent Obstruction vs Late Obstruction vs Persistent Normal; Is there a difference in airway wall thickness among the 4 groups?; Test type: Superiority or Other; p = 0.2, ANOVA

2. Secondary Outcome: Protease/Antiprotease
Description: MMP9/TIMP 1 molar ratio MMP9 is matrix metalloproteinse 9 and is a protease enzyme that is responsible for tissue degradation of extracellular matrix and could be a factor in airway remodeling.
  TIMP 1 is an abbreviation for tissue inhibitor of metalloproteinase-1 and is an inhibitor of MMP9 and would serve to balance the activity protease activity of MMP9 and this it is an anti-protease.
  Therefore the ratio of MMP9 and TIMP1 is used to assess the relative balance of protease and antiprotease activity.
Time Frame: Measured at Year 2
Population: 54 participants had induced sputum data but 1 was excluded due to congenital anatomical anomaly (bronchial atresia).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Persistent Obstruction | Late Obstruction | Late Normal | Persistent Normal
Number analyzed (Participants) | 19 | 7 | 9 | 18
ratio | 34.1 (58.8) | 29.3 (31.3) | 9.9 (8.4) | 12.1 (9.0)

ADVERSE EVENTS:
Arm/Group | Persistent Obstruction | Late Obstruction in Pulmonary Physiology | Late Normal in Pulmonary Physiology | Persistent Normal in Pulmonary Physiology
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/7 | 0/9 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/7 | 0/9 | 0/18

LIMITATIONS AND CAVEATS:
We had planned to extend invitations to the remaining 55 participants in a streamlined version of this protocol after analyzing the preliminary data and an additional cycle of CAMP was funded in 2007.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No